CLINICAL TRIAL: NCT01582698
Title: Open-label Phase 4 Study to Investigate the Seropersistence of Tick-borne Encephalitis (TBE) Virus Antibodies From 7 to 10 Years After the First Booster and the Response to a Second Booster Vaccination With FSME-IMMUN 0.5ml in Adults
Brief Title: TBE Seropersistence up to 10 Years After First Booster in Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 691101; 2011-005557-31 (EudraCT Number); B9371010 (Other: Pfizer)
Record Dates: First submitted 2012-04-20; First posted 2012-04-23 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Tick-borne Encephalitis (TBE)
MeSH Terms: conditions — Encephalitis, Tick-Borne

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Seropersistence evaluation + 2nd booster vaccination (Experimental): Blood will be drawn to assess the seropersistence of TBE virus antibodies at 82, 94, 106 and 118 months after the first booster vaccination with FSME-IMMUN 0.5ml administered during the first precursor study. Timing of the second booster vaccination will depend on the level of serum TBE antibodies observed during the study. Blood will be drawn 21 - 35 days after vaccination to assess the booster response.
  Interventions: Biological: FSME-IMMUN 0.5 ml

INTERVENTIONS:
Biological: FSME-IMMUN 0.5 ml — Solution/suspension for injection (intramuscular injection into the deltoid muscle of the right or left upper arm). Dosage frequency of booster vaccination: dependent on serum TBE antibodies.

SUMMARY:
The purpose of this study is to evaluate TBE antibody persistence from 7 to 10 years after the first booster TBE vaccination with FSME-IMMUN 0.5ml.

ELIGIBILITY:
Inclusion Criteria:

Subjects who participated in the first and second precursor studies will be eligible for participation in this study if:

* they understand the nature of the study, agree to its provisions and provide written informed consent
* they received the first booster vaccination with FSME-IMMUN 0.5ml during the first precursor study and did not receive a second booster vaccination in the second precursor study
* blood was drawn after their first booster vaccination in the first precursor study

Exclusion Criteria:

Subjects will be excluded from participation in this study if they:

* received any TBE vaccination since their first booster vaccination with FSME-IMMUN 0.5ml
* have a history of infection with or vaccination against other flaviviruses (e.g. dengue fever, yellow fever, Japanese B-encephalitis) since their first booster vaccination with FSME-IMMUN 0.5ml
* are known to be HIV positive since their first booster vaccination with FSME-IMMUN 0.5ml
* have a known or suspected problem with drug or alcohol abuse

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2012-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Seropositivity rate measured by neutralization test (NT) 82, 94, 106 and 118 months after the first booster TBE vaccination administered in the first precursor study and after the booster vaccination in this study | 118 months

SECONDARY OUTCOMES:
Seropositivity rate measured by ELISA test 82, 94, 106 and 118 months after the first booster TBE vaccination administered in the first precursor study and after the booster vaccination in this study | 118 months
Antibody titers 82, 94, 106 and 118 months after the first booster TBE vaccination administered in the first precursor study and after the booster vaccination in this study measured by ELISA and by NT | 118 months
Fold increase in antibody concentration after the booster vaccination administered as compared to before the booster vaccination in this study measured by ELISA and by NT | 118 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Poland (2):
  - Prywatny Gabinet Lekarski, Dębica
  - "John Paul II" Cracow Specialist Hospital, Department of Pediatric Neuroinfections and Neurology, Krakow

REFERENCES:
- [Derived] Konior R, Brzostek J, Poellabauer EM, Jiang Q, Harper L, Erber W. Seropersistence of TBE virus antibodies 10 years after first booster vaccination and response to a second booster vaccination with FSME-IMMUN 0.5mL in adults. Vaccine. 2017 Jun 16;35(28):3607-3613. doi: 10.1016/j.vaccine.2017.03.059. Epub 2017 May 22. PMID 28545923